CLINICAL TRIAL: NCT04488081
Title: I-SPY COVID TRIAL: An Adaptive Platform Trial to Reduce Mortality and Ventilator Requirements for Critically Ill Patients
Brief Title: I-SPY COVID-19 TRIAL: An Adaptive Platform Trial for Critically Ill Patients
Acronym: I-SPY_COVID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: QuantumLeap Healthcare Collaborative (Other)
Collaborators: University of California, San Francisco (Other); University of Pennsylvania (Other); Emory University (Other); University of Alabama at Birmingham (Other); University of Colorado, Denver (Other); University of Southern California (Other); Yale University (Other); Wake Forest University Health Sciences (Other); Sanford Health (Other); Long Beach Memorial Medical Center (Other); Georgetown University (Other); University of California, Davis (Other); Hoag Memorial Hospital Presbyterian (Other); Main Line Health (Other); DHR Health Institute for Research and Development (Other); University of California, Irvine (Other); Corewell Health (Unknown); Kaiser Permanente (Other); University of Michigan (Other); West Virginia University (Other); University of Miami (Other); University Hospitals Cleveland Medical Center (Other); Virtua Health (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-SPY-COVID
Record Dates: First submitted 2020-07-14; First posted 2020-07-27 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: COVID-19; severe disease; Platform Trial; Acute Respiratory Distress Syndrome; ARDS; SARS-COV-2; AHRF; Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — COVID-19; Disease; Respiratory Distress Syndrome; Respiratory Insufficiency | interventions — remdesivir; Imatinib Mesylate; Dexamethasone; cenicriviroc; icatibant; apremilast; dornase alfa; Celecoxib; Famotidine; aviptadil; narsoplimab; Cyproheptadine; Cyclosporine

STUDY DESIGN:
Intervention Model Description: Platform Trial, Bayesian Design, from 2 arms up to 8 arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Control/Backbone - Remdesivir and Dexamethasone (CLOSED) (Active Comparator): Participants randomized to the backbone control will be given standard of care (supportive care for ARDS, including remdesivir and, if needed, lung protective ventilation). Because dexamethasone was shown to have benefit in at least one large randomized clinical trial, patients in the backbone control arm should receive dexamethasone for a total of 10 days during the hospitalization or until or hospital discharge.
  Remdesivir (intravenous): 200-mg loading dose on day 1, followed by a daily maintenance dose of 100-mg on days 2 through 10.
  Dexamethasone (intravenous): 6 mg intravenous or oral dexamethasone once daily up to 10 days or equivalent for alternate corticosteroid if dexamethasone unavailable.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone
- Imatinib + Standard of Care (CLOSED) (Experimental): Subjects will be administered standard of care + 800 mg imatinib on Day 1 orally, in divided doses of 400 mg administered twice per day. 400 mg daily will be administered orally for the following 9 days or until discharge, whichever is sooner.
  Interventions: Drug: Remdesivir; Drug: Imatinib Mesylate; Drug: Dexamethasone
- Cenicriviroc + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + cenicriviroc orally , loading 300 mg qAM followed by 150 mg qPM, 12 hours apart on day 1, then 150 mg BID for total of 14 to 28 days depending on date of hospital discharge.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Cenicriviroc
- Icatibant + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + icatibant subcutaneously, a safety run-in for the first 10 subjects was conducted using a regimen of 30 mg q8h × 3 days. All subsequent subjects received drug at 30 mg q8h x 6 days.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Icatibant
- Apremilast + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + apremilast orally , 30 mg bid × 14 days.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Apremilast
- Dornase + Standard of Care (CLOSED) (Experimental): For Non-intubated subjects: Subjects administered standard of care + dornase, 2.5 mg BID until hospital discharge, improvement to room air (or baseline oxygen use prior to illness) for 24 hours, or total of 14 days of study drug, whichever comes first.
  For intubated subjects: Subjects administered standard of care + dornase, 5.0 mg BID in 10 mL normal saline until extubation or 14 days, whichever comes first. If intubated for less than 14 days, extubated subjects received 2.5 mg BID for a total Dornase treatment of 14 days, or until hospital discharge, whichever comes first.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Biological: dornase alfa
- Celecoxib/famotidine + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + celecoxib/famotidine orally .
  Celecoxib, oral: 400 mg BID for 7 days.
  Famotidine, oral: High dose 80 mg QID for 7 days followed by 40 mg BID for a course of 14 days.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Celecoxib; Drug: Famotidine
- IC14 + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + IC14 intravenously , 4 mg/kg on day 1, followed by 2 mg/kg on days 2, 3, 4
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Biological: IC14
- Narsoplimab + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + narsoplimab dosed at 4 mg/kg, given as a 30-minute intravenous infusion (up to a maximum of 370 mg per infusion) twice weekly for a total of four weeks (i.e. 9 doses) or until hospital discharge whichever comes first.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Biological: narsoplimab
- Aviptadil + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + aviptadil (inhalation via nebulizer), 100 µg three times (TID) daily for a maximum of 14 days
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Aviptadil
- Cyproheptadine + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + cyproheptadine via 4 mg tablet, with dosing regimen of 8 mg every 8 hours daily for ten (10) days.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Cyproheptadine
- Cyclosporine + Standard of Care (CLOSED) (Experimental): Subjects administered standard of care + modified cyclosporine at an oral dose of 5mg/kg per day administered in two divided doses daily for 5-days.
  Interventions: Drug: Remdesivir; Drug: Dexamethasone; Drug: Cyclosporine
- Imatinib (PENDING ACTIVATION) (Experimental): Subjects will be administered 800 mg on Day 1 orally, in divided doses of 400 mg administered twice per day. 400 mg daily will be administered orally for the following 9 days or until discharge, whichever is sooner.
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Remdesivir — Participants who receive remdesivir as part of their standard of care will be administered remdesivir by IV for up to ten days. Remdesivir 200mg loading dose on day 1, followed by 100mg IV once daily maintenance doses for 4 or 9 days.
  Other Names: GS-5734
  Arms: Apremilast + Standard of Care (CLOSED); Aviptadil + Standard of Care (CLOSED); Celecoxib/famotidine + Standard of Care (CLOSED); Cenicriviroc + Standard of Care (CLOSED); Control/Backbone - Remdesivir and Dexamethasone (CLOSED); Cyclosporine + Standard of Care (CLOSED); Cyproheptadine + Standard of Care (CLOSED); Dornase + Standard of Care (CLOSED); IC14 + Standard of Care (CLOSED); Icatibant + Standard of Care (CLOSED); Imatinib + Standard of Care (CLOSED); Narsoplimab + Standard of Care (CLOSED)
Drug: Imatinib Mesylate — Subjects will be administered 800 mg on Day 1 orally, in divided doses of 400 mg administered twice per day. 400 mg daily will be administered orally for the following 9 days or until discharge, whichever is sooner.
  Arms: Imatinib (PENDING ACTIVATION); Imatinib + Standard of Care (CLOSED)
Drug: Dexamethasone — 6 mg intravenous of oral dexamethasone once daily up to 10 days or equivalent for alternate corticosteroid if dexamethasone unavailable.
  Arms: Apremilast + Standard of Care (CLOSED); Aviptadil + Standard of Care (CLOSED); Celecoxib/famotidine + Standard of Care (CLOSED); Cenicriviroc + Standard of Care (CLOSED); Control/Backbone - Remdesivir and Dexamethasone (CLOSED); Cyclosporine + Standard of Care (CLOSED); Cyproheptadine + Standard of Care (CLOSED); Dornase + Standard of Care (CLOSED); IC14 + Standard of Care (CLOSED); Icatibant + Standard of Care (CLOSED); Imatinib + Standard of Care (CLOSED); Narsoplimab + Standard of Care (CLOSED)
Drug: Cenicriviroc — Oral, loading 300 mg qAM followed by 150 mg qPM, 12 hours apart on day 1, then 150 mg BID for total of 14 to 28 days depending on date of hospital discharge.
  Arms: Cenicriviroc + Standard of Care (CLOSED)
Drug: Icatibant — Subcutaneous, a safety run-in for the first 10 subjects was conducted using a regimen of 30 mg q8h × 3 days. All subsequent subjects received drug at 30 mg q8h x 6 days.
  Other Names: Firazyr
  Arms: Icatibant + Standard of Care (CLOSED)
Drug: Apremilast — oral, 30 mg bid × 14 days.
  Other Names: Otezla
  Arms: Apremilast + Standard of Care (CLOSED)
Biological: dornase alfa — For Non-intubated subjects: 2.5 mg BID until hospital discharge, improvement to room air (or baseline oxygen use prior to illness) for 24 hours, or total of 14 days of study drug, whichever comes first.
  For intubated subjects: 5.0 mg BID in 10 mL normal saline until extubation or 14 days, whichever comes first. If intubated for less than 14 days, extubated subjects received 2.5 mg BID for a total Dornase treatment of 14 days, or until hospital discharge, whichever comes first.
  Other Names: Pulmozyme
  Arms: Dornase + Standard of Care (CLOSED)
Drug: Celecoxib — Oral: 400 mg BID for 7 days.
  Other Names: celebrex
  Arms: Celecoxib/famotidine + Standard of Care (CLOSED)
Drug: Famotidine — Oral: High dose 80 mg QID for 7 days followed by 40 mg BID for a course of 14 days.
  Other Names: Pepcid
  Arms: Celecoxib/famotidine + Standard of Care (CLOSED)
Biological: IC14 — intravenous, 4 mg/kg on day 1, followed by 2 mg/kg on days 2, 3, 4
  Arms: IC14 + Standard of Care (CLOSED)
Drug: Aviptadil — Inhalation via nebulizer, 100 µg three times (TID) daily for a maximum of 14 days
  Other Names: Zyesami
  Arms: Aviptadil + Standard of Care (CLOSED)
Biological: narsoplimab — Dosed at 4 mg/kg, given as a 30-minute intravenous infusion (up to a maximum of 370 mg per infusion) twice weekly for a total of four weeks (i.e. 9 doses) or until hospital discharge whichever comes first.
  Other Names: OMS721
  Arms: Narsoplimab + Standard of Care (CLOSED)
Drug: Cyproheptadine — 4 mg tablet, with dosing regimen of 8 mg every 8 hours daily for ten (10) days. If the patient weighs less than 48 kg, the regimen is 6 mg every 8 hours daily for ten (10) days. If the participant was discharged before completion of this dosing regimen the drug was not continued.
  Other Names: periactin
  Arms: Cyproheptadine + Standard of Care (CLOSED)
Drug: Cyclosporine — Modified CsA at an oral dose of 5mg/kg per day administered in two divided doses daily for 5-days.
  Other Names: CsA
  Arms: Cyclosporine + Standard of Care (CLOSED)

SUMMARY:
The goal of this project is to rapidly screen promising agents, in the setting of an adaptive platform trial, for treatment of critically ill COVID-19 patients. In this phase 2 platform design, agents will be identified with a signal suggesting a big impact on reducing mortality and the need for, as well as duration, of mechanical ventilation.

DETAILED DESCRIPTION:
This platform trial will provide access to repurposed and investigational agents for critically ill patients infected with SARS-CoV-2 who have severe or life-threatening COVID-19. The main focus of this trial is a platform study for identifying effective agents for the treatment of COVID-19. Any critically ill patient with known or presumed COVID-19 will be automatically entered into the screening phase of the trial until SARS-CoV-2 infection is confirmed. Basic data will be assembled for each patient (such as ventilatory status and survival). If interested in the therapeutic portion of the trial, potential participants will be asked to sign a consent form describing the backbone treatment and the two specific investigational agent arms to which they may be randomized. The primary endpoints will be time to recover to a durable level 4 (or less) on the WHO COVID-19 ordinal scale for clinical improvement and time to mortality (death). For this trial, a durable level 4 is defined as at least 48 hours at COVID level 4 or less (nasal prongs oxygen) without returning to high flow oxygen or intubation. Acute care facility resource utilization will be automatically calculated (total length of stay in a critical care setting, days intubated, and survival). Any change in status, including intubation, extubation, death or discharge, will be recorded and verified by the attending physician.

Patients will be evaluated based on their initial status (ventilation at entry vs. high flow oxygen). Exploratory biomarkers will be evaluated over time (ARDS phenotypes and other proposed markers) to facilitate clinical learning. A maximum of two investigational arms may be open at a time. The anticipated accrual will be 50 patients per week. The maximum number of participants assigned to an arm without graduation will be 125 patients. Agents can be dropped for futility after enrollment of 40 patients. As the trial proceeds and a better understanding of the underlying mechanisms of the COVID-19 illness emerges, expanded biomarker and data collection can be added as needed to further elucidate how agents are or are not working. The study design features comparison of investigational agent efficacy using a Bayesian design, which will allow the detection of strong efficacy signals with the fewest possible patients. Initially the control will be patients given current standard of care (supportive care for ARDS, including lung protective ventilation and remdesivir and dexamethasone as backbone therapy). As other treatments (for example, anticoagulation) become part of standard supportive care across sites, these will be added to the backbone therapy. If an agent meets the threshold for graduation the company leadership will be informed as will the FDA. The arm with the graduated agent will cease to enroll, allowing a new arm with a different investigational agent to be added.

Every trial participant will have blood collected at trial enrollment, day 3, and day 7 for pre-specified biomarker and DNA and RNA analysis. Additional biomarkers can be added as the trial proceeds. Patient outcomes will also be evaluated on the basis of whether patients are ventilated initially or not.

Observational Component:

Initially, all COVID-19 confirmed patients who started high-flow oxygen (WHO COVID-19 level 5; ≥6L oxygen by nasal prongs or mask) were entered in an Observational Component which collected data via extraction of medical records. Patients in this Observational Component also had their daily COVID status and drug administration form CRFs completed. An expanded Observational Study will replace the original Observational Component. The expanded observational study (Supplement 1) will collect blood sample(s) and clinical data from ARDS and AHRF patients (including COVID ARDS patients) to test the feasibility of quantifying a set of biomarkers that will allow each patient to be classified into either a hyper-inflammatory or hypo-inflammatory subtype in real time. If treatment of these critically ill ICU patients is to be guided by subtype classification, it is essential that the operational time for classification is as quick as possible.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

A. Male or Female, at least 18 years old

B. Admitted to the hospital and placed on high flow oxygen (≥6L by nasal cannula or mask delivery system) or intubated for the treatment of (established or presumed) COVID-19.

C. Informed consent provided by the patient, LAR or health care proxy.

D. Confirmation of SARS-CoV-2 infection by PCR or Rapid antigen testing for SARS- CoV-2 infection prior to randomization.

Exclusion Criteria:

A. Pregnant or breastfeeding women (must be documented by a pregnancy test during hospitalization)

B. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent based on review of the medical record and patient history.

C. Comfort measures only.

D. Acute liver disease, or chronic liver disease with a Child-Pugh score greater than 11.

E. Resident for more than six months at a skilled nursing facility.

F. Estimated mortality greater than 50% over the next six months from underlying chronic conditions.

G. Time since requirement for high flow oxygen or ventilation greater than 5 days.

H. Anticipated transfer to another hospital which is not a study site within 72 hours.

I. Patients with either end-stage kidney disease or acute kidney injury who are on dialysis.

J. Co-enrollment in clinical trials of pharmacologic agents requiring an IND.

K. On 3 or more vasopressors.

L. Pre-existing heart failure with a known left ventricular ejection fraction <25% or unstable angina pectoris.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-07-31 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Identify agents that will result in substantial improvements to the clinical condition of participants with COVID-19. | Up to 28 days
  Time to reach a durable COVID-19 level 4 or less or discharge at COVID-level 4 or lower (except for discharge to another hospital), and time to death (mortality).
  Data will be analyzed for 3 groups:
  * All
  * COVID-19 level 6/7 (those intubated immediately)
  * COVID-19 level 5 (high flow oxygen to start)
  World Health Organization 9-point ordinal scale:
  0. No clinical or virologic evidence of infection
  1. Not hospitalized, no limitations on activities;
  2. Not hospitalized, limitation on activities;
  3. Hospitalized, not requiring supplemental oxygen;
  4. Hospitalized, requiring supplemental oxygen (< 6L by nasal cannula or mask delivery system);
  5. Hospitalized, on non-invasive ventilation or high flow oxygen devices (≥6L per minute, mask or intranasal cannula);
  6. Hospitalized, on invasive mechanical ventilation;
  7. Hospitalized, ventilation plus additional organ support-pressors, RRT, ECMO
  8. Death.

SECONDARY OUTCOMES:
Mortality | Up to 28 days
  * Proportion of patients alive in the treatment and control arm at day 7, 14, 21, and 28 (The proportion of patients alive, i.e., alive and still at risk of both reaching level 4 and death is given by the survival function).
  * The cumulative incidence function for mortality.
Improvement in disease severity | Up to 60 days
  * Sustained recovery which is defined as time to discharge at COVID-level 4 or lower and not subsequently re-admitted to the hospital or die at Day 28 follow-up if discharged before 28 days, and Day 60 follow-up if discharged between 28 to 60 days.
  * % of COVID-19 level 5 who never progress to COVID-19 level 6/7
  The measure for recovery is defined as time to reach level 4 or less in the World Health Organization COVID-19 scale for at least 48 hours - without returning to high flow oxygen or intubation, or discharge at COVID level 4 or less except for discharge to another hospital. (0 being minimum and 8 being maximum)
Health care utilization | Up to 28 days
  Ventilator-free days
Safety: Frequency of serious AEs | Up to 60 days
  * Total grade 3 or higher AEs by arm and total number of patients with grade 3 or higher AEs by arm.
  * Total grade 3 or higher AEs of special interest by arm and total number of patients with grade 3 or higher AEs of special interest by arms (based upon lab assessments)
  All AEs will be identified and assessed for severity using the National Cancer Institute - Common Terminology Criteria for Adverse Events v5.0 which provides a grading scale for each AE listed.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL*.
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL**.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Carolyn, MD, Principal Investigator — University of California, San Francisco; Kathleen D Liu, MD, Principal Investigator — University of California, San Francisco; Laura Esserman, MD, Principal Investigator — University of California, San Francisco
Locations (36):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Davis Medical Center, Davis, California
  - UC Irvine Medical Center, Irvine, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Kaiser LAMC, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - University of California San Francisco (UCSF), San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Stamford Health, Stamford, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Mercy Hospital Springfield, Springfield, Missouri
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Virtua Mount Holly Hospital, Mount Holly, New Jersey
  - Virtua Voorhees Hospital, Voorhees Township, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania (U Penn), Philadelphia, Pennsylvania
  - Lankenau Medical Center (Mainline Health), Wynnewood, Pennsylvania
  - Main Line Health - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - DHR Health, Edinburg, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - WVU Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
We will share data on a case by case basis with appropriate IRB review and review by our Data Safety Monitoring Comittee.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Post publication or earlier if warranted.
Access Criteria: Sharing criteria are based on the circumstances of the request and whether the data have been published.

REFERENCES:
- [Background] Files DC, Matthay MA, Calfee CS, Aggarwal NR, Asare AL, Beitler JR, Berger PA, Burnham EL, Cimino G, Coleman MH, Crippa A, Discacciati A, Gandotra S, Gibbs KW, Henderson PT, Ittner CAG, Jauregui A, Khan KT, Koff JL, Lang J, LaRose M, Levitt J, Lu R, McKeehan JD, Meyer NJ, Russell DW, Thomas KW, Eklund M, Esserman LJ, Liu KD; ISPY COVID Adaptive Platform Trial Network; undefined. I-SPY COVID adaptive platform trial for COVID-19 acute respiratory failure: rationale, design and operations. BMJ Open. 2022 Jun 6;12(6):e060664. doi: 10.1136/bmjopen-2021-060664. PMID 35667714
- [Derived] Mabrey FL, Martin TR, Calfee CS, Liu KD, LaCombe B, Brown-Swigart L, Discacciati A, Eklund M, Heckbert SR, Matthay MA, Esserman L, Wurfel MM. Anti-CD14 treatment in patients with severe COVID-19: Clinical and biological effects in a Phase 2 randomized open-label adaptive platform clinical trial. CHEST Crit Care. 2025 Mar;3(1):100117. doi: 10.1016/j.chstcc.2024.100117. Epub 2024 Dec 9. PMID 40462830
- [Derived] Pomponio R, Peterson RA, Owusu M, Slaughter S, Melgar S, Jolley SE, Burnham EL. Phosphatidylethanol measures in patients with severe COVID-19-associated respiratory failure identify a subset with alcohol misuse. Alcohol Clin Exp Res (Hoboken). 2025 Jan;49(1):165-174. doi: 10.1111/acer.15495. Epub 2024 Nov 26. PMID 39592213
- [Derived] I-SPY COVID Consortium. Report of the first seven agents in the I-SPY COVID trial: a phase 2, open label, adaptive platform randomised controlled trial. EClinicalMedicine. 2023 Apr;58:101889. doi: 10.1016/j.eclinm.2023.101889. Epub 2023 Mar 3. PMID 36883141
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: Clinical trial design during and beyond the pandemic: the I-SPY COVID trial, 20Jan2022 — https://www.nature.com/articles/s41591-021-01617-x